CLINICAL TRIAL: NCT03904186
Title: Effectiveness of an Integrated Treatment to Address Smoking Cessation and Anxiety/ Depression in People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Fenway Institute (Other); University of Texas at Austin (Other); University of Houston (Other); Baylor College of Medicine (Other); Southern Methodist University (Other)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Associate Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA047933 (NIH)
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Human Immunodeficiency Virus; Smoking Cessation; Smoking, Cigarette; Smoking; Anxiety; Depression; Nicotine Dependence
Keywords: Tobacco Use; Tobacco Use Disorder; Substance-Related Disorders; Nicotine; Ganglionic Stimulants; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Nicotinic Agonists; Cholinergic Agonists; Cholinergic Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; HIV; Anxious; Anxiety Symptoms; Depressive Symptoms; Quitting; Cognitive Behavioral Therapy; Anxiety Sensitivity; Distress Intolerance; Anhedonia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking Cessation; Cigarette Smoking; Smoking; Anxiety Disorders; Depression; Tobacco Use Disorder; Tobacco Use; Substance-Related Disorders; Anhedonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QUIT Treatment for Smoking Cessation and Distress Tolerance (Experimental): Participants in this intervention arm will receive a Cognitive-Behavioral therapy-based intervention for smoking cessation in people living with HIV.
  Interventions: Behavioral: QUIT
- Time and Intensity-Match Control (Active Comparator): Participants in this control arm will receive an intervention matched in time and intensity with the experimental arm.
  Interventions: Behavioral: Time-Matched Control (TM)
- Standard of Care (No Intervention): At each clinic, routine assessment of smoking status occurs at least annually for patients receiving care, but prescription for pharmacotherapy for smoking cessation and referral for behavioral smoking cessation services are rare. Patients will receive the standard of care at the clinic they attend. SOC patients will also attend the first session that participants in the other sessions receive (pre-randomization), will come to the clinic for assessment only during the weeks lining up with sessions 6-10 for the other conditions, and receive the transdermal nicotine patch for 8 weeks.

INTERVENTIONS:
Behavioral: QUIT — QUIT is a transdiagnostic Cognitive Behavioral Therapy-based smoking cessation protocol designed to address distress intolerance, anxiety sensitivity, and anhedonia in people living with HIV who smoke. QUIT is delivered in 9 60-minute individual weekly sessions over a 10-week period. Sessions are active, with treatment components practiced within and outside of the session. Participants will also receive the transdermal nicotine patch for 8 weeks, starting when they attempt to quit smoking during week 7 of the study.
  Arms: QUIT Treatment for Smoking Cessation and Distress Tolerance
Behavioral: Time-Matched Control (TM) — Participants will receive a standard smoking cessation treatment, based on the clinical practice guidelines from the U.S. Department of Health and Human Services, Treating Tobacco Use and Dependence. Treatment will be delivered in nine, 60-minute sessions over a ten-week period. The treatment is based on a treatment protocol developed and used previously by Dr. Zvolensky. Because clinical guidelines recommend that all smokers attempting to quit smoking receive pharmacotherapy, participants will also receive the transdermal nicotine patch for 8 weeks.
  Arms: Time and Intensity-Match Control

SUMMARY:
Smokers living with HIV represent a major health disparity population in the United States and the world more generally. Major contributing factors to the maintenance and relapse of smoking among smokers living with HIV include increased exposure to multiple stressors associated with HIV, which often exacerbates anxiety/depression. In a previous project, the feasibility, acceptability, and initial efficacy of a 9-session, cognitive-behavioral-based intervention to address smoking cessation by reducing anxiety and depression via specific emotional vulnerabilities (anxiety sensitivity, distress tolerance, and anhedonia) was tested against an enhanced standard of care in a pilot randomized controlled trial (NCT01393301). It was found that when compared to a brief enhanced treatment as usual control, patients in the intervention achieved higher short-term and long-term smoking abstinence rates. In this project, the investigators seek to test this same intervention in a fully powered, 3-arm efficacy/effectiveness trial. The goal of this study is to randomize 180 smokers across three sites to test the efficacy/effectiveness of the intervention at increasing point prevalence abstinence by reducing anxiety and depression at a 1-month follow-up (the end of treatment timepoint/ approximately 1-month post quit day) and a 6-month follow-up (approximately 6-months post quit day).

DETAILED DESCRIPTION:
Although the prevalence of smoking has declined over the past 50 years, large disparities in tobacco use remain across several subgroups, particularly disadvantaged and health compromised populations. In fact, the initiation and maintenance of smoking is twice as likely for individuals living with HIV than individuals not living with HIV. Smokers living with HIV represent a major health disparity population in the United States (US) and the world more generally, and their unique healthcare needs are not being adequately addressed. For people living with HIV, smoking is related to poorer survival, and among those who are adherent to their antiretroviral treatment regimens, smoking reduces life expectancy more than HIV. A major contributing factor to the maintenance and relapse of smoking among smokers living with HIV is the increased exposure to multiple stressors associated with HIV (e.g., compromised health status, stigma, cognitive impairment), which in turn, contributes to heightened anxiety/depression. Further, smokers living with HIV tend to rely on smoking to regulate their negative mood. As a result, smokers living with HIV require specialty care options that address their unique 'affective needs.' The proposed intervention is informed by the success of a recently completed research project (NCT01393301) in which the feasibility and acceptability of a 9-session, cognitive-behavioral therapy-based intervention to address smoking cessation and symptoms of anxiety and depression by targeting common processes underlying anxiety/depression (distress intolerance, anxiety sensitivity, anhedonia) was tested in a pilot randomized controlled trial (RCT) against an enhanced treatment as usual condition. Investigators named this intervention "QUIT". In the pilot RCT, smoking abstinence was significantly higher in the intervention than in the standard of care control at both the 1-month follow-up (the end-of-treatment timepoint) and the 6-month follow-up, and anxiety and depressive symptom severity was lower in the intervention condition than the control condition at the same timepoints. The present study seeks to conduct a fully powered, 3-arm hybrid efficacy/effectiveness trial, integrating resource utilization and cost-effectiveness analyses. The investigators propose to randomize 180 smokers living with HIV across three implementation sites. Two-fifths of the sample (n = 72) will be randomized to the QUIT intervention; two-fifths (n = 72) to an active, credible time-matched control (TM) and one-fifth (n = 36) to a standard-of-care (SOC) control. The primary outcomes of this study will be point prevalence abstinence at the 1-Month Follow-Up (end of treatment timepoint/ approximately 1-month post quit day) and 6-Month Follow-Up (approximately 6-months post quit day). Changes in anxiety/depressive symptom severity will also be examined, and cost-effectiveness analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18-79 years old
* Daily Smoker
* Motivated to quit smoking
* HIV-positive
* Capability and willingness to give written informed consent

Exclusion Criteria:

* Habitual use of tobacco products other than cigarettes
* Untreated or unstable psychiatric disorders
* Current smoking cessation treatment
* Cognitive behavioral therapy for anxiety within the past year
* Insufficient command of the English language

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Short-Term Point Prevalence Smoking Abstinence | Time frame: 1-Month Follow-Up (end of treatment/approximately 1-month post quit date)
  Biologically verified 7-day point prevalence abstinence (PPA). Using the timeline follow-back method (TLFB), participants will self-report the last time they smoked. TLFB results will be biologically verified with carbon monoxide analysis of breath samples (if stated abstinence is between 24 hours and 2 weeks), saliva cotinine (if stated abstinence is 2+ weeks and participant is currently using nicotine replacement therapy), or urine anabasine (if stated abstinence is 2+ weeks and participant is not currently using nicotine replacement therapy).
Long-Term Point Prevalence Smoking Abstinence | Time frame: 6-Month Follow-Up (approximately 6-months post quit date)
  Biologically verified 7-day point prevalence abstinence (PPA). Using the timeline follow-back method (TLFB), participants will self-report the last time they smoked. TLFB results will be biologically verified with carbon monoxide analysis of breath samples (if stated abstinence is between 24 hours and 2 weeks), saliva cotinine (if stated abstinence is 2+ weeks and participant is currently using nicotine replacement therapy), or urine anabasine (if stated abstinence is 2+ weeks and participant is not currently using nicotine replacement therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, PhD, Principal Investigator — University of Texas at Austin; Michael Zvolensky, PhD, Principal Investigator — University of Houston
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fenway Community Health, Boston, Massachusetts
  - Thomas Street Health Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
One year following achievement of aims of the project (i.e., publication of the main outcome paper), de-identified data from this project will be provided to interested individuals. These data will be provided in digital format with clear labels for all variables. Data will be released directly by the investigators providing evidence of their institution's IRB approval for planned analyses of the data. The study team will be available to address queries.

REFERENCES:
- [Derived] Garey L, Wirtz MR, Labbe AK, Zvolensky MJ, Smits JAJ, Giordano TP, Rosenfield D, Robbins GK, Levy DE, McKetchnie SM, Bell T, O'Cleirigh C. Evaluation of an integrated treatment to address smoking cessation and anxiety/depressive symptoms among people living with HIV: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2021 Jul;106:106420. doi: 10.1016/j.cct.2021.106420. Epub 2021 Apr 30. PMID 33933667